CLINICAL TRIAL: NCT03695523
Title: Examining a Childcare Policy to Promote Physical Activity Among Young Children
Brief Title: PLAY (PhysicaL ActivitY) Policy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 111890; 43670 (Other Grant/Funding Number: WSS-MHSRB Accelerator Grant)
Record Dates: First submitted 2018-09-18; First posted 2018-10-04 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2018-08

CONDITIONS: Motor Activity
Keywords: Physical activity; Children; Child care; Policy; Accelerometer
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Children and childcare providers will be aware of whether or not they receive the intervention. However, research assistants who are collecting data will remain blind to each centre's group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PLAY (PhysicaL ActivitY) Policy Intervention (Experimental): The childcare physical activity policy will be adopted for 8 weeks within participating toddler and preschool classrooms of facilities allocated to the experimental group.
  Interventions: Behavioral: PLAY (PhysicaL ActivitY) Policy Intervention
- Control group (No Intervention): Childcare centres will maintain their typical daily programming and standard of care for the duration of the 8-week intervention period.

INTERVENTIONS:
Behavioral: PLAY (PhysicaL ActivitY) Policy Intervention — An evidence-based physical activity policy that was developed by researchers and childcare stakeholders and directed by the Canadian 24-Hour Movement Guidelines for the Early Years will be adopted by experimental group childcare centres for 8 weeks. The policy incorporates 8 items (i.e., encouraging children to engage in higher intensity energetic play often, aiming to accumulate 40 minutes each day, exposing children to a variety of indoor and outdoor physical activities, child-directed and teacher-facilitated active play daily, short bouts of outdoor time for a total of 120 minutes each day made up of primarily unstructured free play, encouraging physical literacy by practicing fundamental movement skills, not exposing children to screen-based technology during childcare, and purposefully breaking up sustained sedentary time using physical activities).
  Other Names: Examining a childcare policy to promote children's physical activity
  Arms: PLAY (PhysicaL ActivitY) Policy Intervention

SUMMARY:
This study examines the effectiveness and appropriateness of a written physical activity policy implemented in licensed centre-based childcare on the physical activity levels of toddlers (1-2) and preschoolers (3-5 years). Half of the childcare centres will adopt the physical activity policy while the other half will continue with their typical daily programming and care. It is hypothesized that children enrolled in childcare centres that adopt the policy will display increased levels of physical activity during, and after participating in the policy intervention compared to children enrolled in centres that do not adopt the policy.

DETAILED DESCRIPTION:
A pilot, cluster single-blind randomized controlled trial (RCT) will be conducted. Approximately 8 licensed childcare centres will be randomly selected from an online listing of centres in London, Canada. Since it is necessary to implement the policy at the centre-level to groups of children, the childcare centres (i.e., the clusters) rather than the individual participants, will be randomly allocated to either implement the physical activity policy (experimental; n = 4), or maintain their daily programming (control; n = 4) for the 8-week intervention period.

In both groups, toddlers' and preschoolers' physical activity will be objectively measured using motion sensors (ActiGraph wGT3X-BT accelerometers) worn on an elastic waistband for 5 consecutive days, during childcare hours, before the policy is implemented (baseline; week 0; September 2018), mid-intervention (week 4; October 2018), one week after the intervention period ends (post-intervention; week 9; November/December 2018), and 6-months post-intervention (May-June 2019).

The aim of the study is to examine the impact of a childcare physical activity policy on the objectively measured physical activity levels (light physical activity, LPA; moderate-to-vigorous physical activity, MVPA), and combined total physical activity (TPA), and sedentary time of young children in childcare centres compared to children from centres that maintain their usual standard of care.

ELIGIBILITY:
Inclusion Criteria:

For childcare centres:

* Must be a licensed centre-based childcare facility in London, Ontario, Canada or surrounding area
* Must provide care to toddlers and/or preschoolers and must have at least one toddler or preschool-age classroom
* Must have childcare providers in these classrooms who are willing to participate
* Must speak and read English
* Must not have an institutional-level physical activity policy in place

For childcare providers:

* Must be a full-time childcare provider in a toddler or preschool-age classroom of one of the participating centres
* Must speak and understand English

For toddler/preschool participants:

* Must be enrolled in a classroom of a participating centre
* Must be between the ages of 1-5 years of age at baseline (and therefore enrolled in their toddler or preschool-age classrooms)
* Must be expected to remain in childcare for the next 8 months
* Must have a parent/guardian that can read and write English
* Must speak and understand English
* Must receive parental consent

Exclusion Criteria:

For childcare centres:

* Not be located in London and surrounding area
* Not have a toddler or preschool-age classroom
* No childcare providers in any classroom who are willing to participate
* Not an English-speaking facility
* Already has an established physical activity policy in place

For childcare providers:

* Not full time
* Not a childcare provider in a toddler or preschool age classroom at a participating centre
* Does not speak/read/write English

For toddler/preschooler participants:

* Not between the ages of 1 and 5 at baseline
* Not expected to remain in childcare for the next 8 months
* Not enrolled in toddler or preschool classroom of a participating centre
* Does not speak English
* Parent/guardian does not read/write in English

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 278 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-06-29 (Actual); Study Completion 2019-06-29 (Actual)

PRIMARY OUTCOMES:
Changes in young children's Total Physical Activity (TPA) | Measured for 5 consecutive days at baseline (i.e., week 0), mid-intervention (i.e., week 4), post-intervention (i.e., week 9), and at 6-months post-intervention.
  TPA, the accumulation of light-, moderate-, and vigorous-intensity physical activity will be assessed using ActiGraph wGT3X-BT accelerometers worn on each child's right hip for 5 consecutive days during childcare hours only at 4 time-points. Differences in TPA will be compared across groups (control vs. experimental) and over time (i.e., week 0, week 4, week 9, and 6 months post-intervention).

SECONDARY OUTCOMES:
Changes in children's Moderate-to-Vigorous Physical Activity (MVPA) | Measured for 5 consecutive days at baseline (i.e., week 0), mid-intervention (i.e., week 4), post-intervention (i.e., week 9), and at 6-months post-intervention.
  Assessed using ActiGraph wGT3X-BT accelerometers worn on each child's right hip for 5 consecutive days during childcare hours only. Differences in MVPA across groups (control vs. experimental) and over time will be assessed.
Changes in children's Sedentary Time (ST) | Measured for 5 consecutive days at baseline (week 0), mid-intervention (week 4), post-intervention (week 9), and at 6-months post-intervention.
  Assessed using ActiGraph wGT3X-BT accelerometers worn on each child's right hip for 5 days during childcare hours only. Differences between groups (control vs. experimental) and across time will be assessed.
Self-efficacy scale for physical activity | Providers will be asked to complete this survey one week prior to baseline measures (Time 1), at baseline (i.e., week 0; Time 2), then again at mid-intervention (i.e., week 4; Time 3), post-intervention (i.e., week 9; Time 4), and at 6 months follow-up.
  Developed for the study to assess childcare providers' self-efficacy to engage children in physical activity during hours of care. Providers are instructed to rate their confidence to each of 40 items on a Likert scale from 1 (no confidence at all) to 5 (somewhat confident) to 10 (completely confident). The psychometric properties of the scale will be evaluated, and childcare providers' self-efficacy may be examined as a correlate of children's objectively measured physical activity. Changes in self-efficacy across groups and time will be assessed.
Environment and Policy Assessment and Observation Self-Report Today (EPAO-SR Today) | Administered to childcare providers in participating classrooms to complete once at baseline (i.e., week 0), mid-intervention (i.e., week 4), post-intervention (i.e., week 9), and at 6-months follow-up.
  Developed and validated by Ward and colleagues (2015), this tool, adapted for use in Canada, without the nutrition scale, provides a snapshot of the daily childcare practices related to physical activity and screen-based sedentary time. Data will be compared across groups (control vs. experimental) and across time (week 0, week 4, week 9, and at 6 months follow-up).
Policy intervention implementation log | Childcare providers within participating classrooms will be asked to complete the log on three days of each week of the 8-week intervention period.
  A self-report log completed by childcare providers in experimental classrooms. Developed for the study to evaluate adherence to the PLAY policy within each classroom.
Director Environment and Policy Assessment and Observation Self-Report (EPAO-SR) | Completed at baseline (i.e., week 0) only.
  Developed and validated by Ward et al. (2015), this tool, adapted for use in Canada without the nutrition scale, measures each centre's physical space, equipment, environment, and existing physical activity policy and practices as reported by directors. This will be used as a screening tool to indicate any physical activity policies already in effect.
Feasibility and appropriateness | Conducted post-intervention (after week 9)
  Focus groups conducted with experimental group childcare providers will provide feedback on the feasibility and appropriateness of the policy. The challenges and solutions used to overcome these challenges will be discussed. Suggestions for potential modifications and improvements to the policy will be collected to inform future iterations for further investigation with larger, more diverse samples.

CONTACTS AND LOCATIONS:
Overall Officials: Trish Tucker, PhD, Principal Investigator — University of Western Ontario, Canada
Locations (1):
- University of Western Ontario - Child Health and Physical Activity Lab, London, Ontario, Canada

REFERENCES:
- [Derived] Szpunar M, Driediger M, Johnson AM, Vanderloo LM, Burke SM, Irwin JD, Shelley J, Timmons BW, Tucker P. Impact of the Childcare Physical Activity (PLAY) Policy on Young Children's Physical Activity and Sedentary Time: A Pilot Clustered Randomized Controlled Trial. Int J Environ Res Public Health. 2021 Jul 13;18(14):7468. doi: 10.3390/ijerph18147468. PMID 34299917